CLINICAL TRIAL: NCT07249996
Title: Respiratory Infections in Young Children in Colombia and Panamá: Epidemiology, Interactions, and Long-term Consequences.
Brief Title: Respiratory Infections in Young Children
Acronym: MINERVAL
Status: Recruiting | Type: Observational
Sponsor: Eduardo Lopez -Medina (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Eduardo Lopez -Medina, Scientific Director, CEIP, Centro de Estudios en Infectogía Pediatrica
Organization: Centro de Estudios en Infectogía Pediatrica (Other)
Other Study IDs: 103600
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Tract Infections (RTI); Lower Respiratory Tract Infection (LRTI); Viral Infections; Cohort Study
Keywords: Birth Cohort Study; Respiratory Tract Infection (RTI); Children
MeSH Terms: conditions — Respiratory Tract Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood Samples, Nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- • Newborns younger than 29 days of life, with or without pre-existing conditions: Infants whose parent(s) or guardian(s) are available for telephone contact for the duration of the study, do not intend to relocate outside of the study area, provide informed consent to participate in the study and are willing to authorize data and specimen collection, storage and analysis.

SUMMARY:
The goal of this observational study is to learn about the causes, severity, and long-term effects of respiratory tract infections (RTIs) in young children from birth to five years of age in Colombia and Panamá. The main questions it aims to answer are:

How often do respiratory infections occur in children under two years old, and which viruses or bacteria cause them? Why do some children develop more severe infections than others? Do early infections or vaccinations change how the immune system responds to future illnesses? How do viruses and bacteria interact in the respiratory tract to influence disease severity and long-term respiratory health? Researchers will follow newborns from birth until age five to understand how respiratory infections develop and affect children's health over time. Participants will not receive any experimental treatment.

Families who join the study will:

Be contacted twice a week through a phone app or phone calls to check for symptoms of respiratory infection.

Attend in-person visits if their child becomes ill and every six months for routine follow-up.

Provide nasal and blood samples during illness episodes so researchers can identify the viruses or bacteria causing infection and study how the immune system responds.

This study began in May 2024 and is being conducted in Cali, Colombia, and Panamá City, Panamá. The research team plans to continue to include participants and continue active follow-up until the children reach five years of age.

The information collected will help scientists and health professionals understand how different pathogens cause respiratory infections, what factors increase the risk of severe illness, and how early infections may influence long-term lung health. The study's findings will support future efforts to prevent and treat respiratory diseases in young children.

DETAILED DESCRIPTION:
Respiratory tract infections (RTIs) remain one of the most common causes of illness and death in young children, despite advances in vaccination and health programs. In children under five years of age, RTIs cause significant morbidity, social costs, and long-term health consequences. The clinical spectrum of RTI ranges from mild upper infections to severe lower respiratory tract infections (LRTIs) such as bronchiolitis and pneumonia. Viruses are the leading cause, especially in the first two years of life. However, in Latin America, there is limited information about how often RTIs occur, what viruses or bacteria are responsible, and how severe these infections are in community settings. Most existing data come from hospitalized cases, which underestimate the real disease burden.

To address this gap, researchers launched the MINERVAL study, a multicenter, prospective birth cohort conducted in Cali, Colombia, and Panamá City, Panamá. The study began in May 2024 and follows children from birth to five years of age to better understand the epidemiology, etiology, and consequences of RTIs. A total of 436 newborns have been enrolled as of February 2025. This population-based cohort is followed by active surveillance twice a week using a phone app or calls, with in-person visits during RTI episodes and routine visits every six months in the first two years of life. From ages two to five, children continue follow-up every six months to assess long-term outcomes.

The study has four main objectives: (1) to determine the incidence, etiology, and seasonality of RTIs in children aged 0-2 years; (2) to assess the pathogen-specific burden of infections caused by viruses such as RSV, hMPV, influenza, SARS-CoV-2, and others across outpatient and inpatient settings; (3) to evaluate long-term respiratory sequelae of LRTIs during early life and their association with chronic respiratory illness by age five; and (4) to analyze viral-bacterial interactions, focusing on how pneumococcal bacterial loads and immune responses influence disease progression.

Preliminary data from 436 participants show 222 RTI episodes, including 42 LRTIs. The cumulative incidence of RTI was 40% at 100 days and 64.8% at 250 days. For LRTIs, incidence was 8.9% at 100 days and 12.2% at 250 days. Among LRTIs, 82.9% were mild, 14.6% moderate, and 2.4% severe. More than half of LRTI episodes required hospitalization, and 14.3% required intensive care. Samples have been collected from 91% of episodes for laboratory analysis.

These findings confirm the feasibility of long-term active surveillance in this cohort and the high frequency of early-life respiratory infections. The continued study will provide critical insights into the incidence, mechanisms, and long-term health consequences of RTIs in Latin American children, supporting the development of new preventive and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Newborns younger than 29 days of life, with or without pre-existing conditions
* Infants whose parent(s) or guardian(s) are available for telephone contact for the duration of the study, and do not intend to relocate outside of the study area, to ensure adherence to RTI and in-person visits.
* Infants whose parent(s) or guardian(s) provide informed consent to participate in the study.
* Infants whose parent(s) or guardian(s) are willing to authorize data and specimen collection, storage and analysis.

Exclusion Criteria:

* Infants born to a pregnant mother under 14 years of age (under Colombian law, pregnancies occurring in individuals younger than 14 years of age are legally presumed to result from sexual abuse).

Max Age: 29 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns younger than 29 days of life, with or without pre-existing conditions
Sampling Method: Non-Probability Sample
Enrollment: 1088 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2031-05-02 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate | From enrollment, up to 2 years of age.
  The number and etiology of new cases of RTI and LRTI according to cumulative time at risk and month of occurrence, in children aged 0 to 2 years.

SECONDARY OUTCOMES:
Severity by pathogen | From enrollment, up to 2 years of age
  Frequency of children who develop RTI, and mild, moderate or severe LRTI, according to pathogen and maximum level of care (outpatient care, emergency room, hospital admission or intensive care) and oxygen support (none, nasal canula, non-invasive ventilation or mechanical ventilation) received by children with LRTI, according to pathogen
Burden in in-patient and outpatient settings | From recruitment, up to 2 years of age
  Median Duration of symptoms, Hospitalization rates, Length of hospital stay, Use of medications, Antibiotic consumption, Lost workdays and daily activities due to illness
Pneumococcal bacterial load and Host immune response | From recruitment, up to 2 years of age
  Disease severity according to pneumococcal bacterial loads and whole blood transcriptome analysis.

OTHER OUTCOMES:
Long term Sequelae | From recruitment to study completion at 5 years
  Prevalence of chronic respiratory illness, recurrent wheezing or asthma, up to 5 years of age, according to the etiology of lower RTI diagnosed during the first two years of life

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Lopez-Medina, MD, MSc, Principal Investigator — Centro de Estudios en Infectologia Pediatrica, CEIP
Locations (2):
- Centro de Estudios en Infectologia Pediatrica, CEIP, Cali, Valle del Cauca Department, Colombia
- Cevaxin, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No